CLINICAL TRIAL: NCT02835339
Title: Randomized Trial of Magnesium Sulfate in Obese Preeclamptic Women
Brief Title: Magnesium Sulfate in Obese Preeclamptics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kathleen Brookfield, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB 15809
Record Dates: First submitted 2016-07-07; First posted 2016-07-18 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MgSO4 4g load, 1g/hr infusion (Active Comparator): Once their obstetrician prescribes magnesium sulfate, participant will be assigned by 50/50 chance to one of two treatment regimens. Participant will be assigned to either a dose of 4 g at the start, followed by 1g every hour; or a dose of 6 g at the start, followed by 2g every hour until treatment for preeclampsia is complete.
  Interventions: Drug: Magnesium sulfate 4g loading dose, 1g/hr infusion
- MgSO4 6g load, 2g/hr infusion (Experimental): Once their obstetrician prescribes magnesium sulfate, participant will be assigned by 50/50 chance to one of two treatment regimens. Participant will be assigned to either a dose of 4 g at the start, followed by 1g every hour; or a dose of 6 g at the start, followed by 2g every hour until treatment for preeclampsia is complete.
  Interventions: Drug: Magnesium sulfate 6g loading dose, 2g/hr infusion

INTERVENTIONS:
Drug: Magnesium sulfate 4g loading dose, 1g/hr infusion
  Arms: MgSO4 4g load, 1g/hr infusion
Drug: Magnesium sulfate 6g loading dose, 2g/hr infusion
  Arms: MgSO4 6g load, 2g/hr infusion

SUMMARY:
The purpose of this study is to learn how medications participant will receive in the course of their delivery are metabolized (broken down by the body). The investigators hope to learn more about the way drugs are metabolized by pregnant women, and how those drugs are distributed in the blood and body compartments and cleared in the urine, and how maternal body weight affects the metabolism. With this information the investigators will be able to develop a treatment regimen considering factors in the body that affect magnesium levels so that the investigators can improve treatment of pregnant women. The goal of the study is to understand how different dosing of magnesium sulfate affects blood levels of the magnesium in larger women.

DETAILED DESCRIPTION:
The purpose of this study is to learn how medications participant will receive in the course of their delivery are metabolized (broken down by the body). The investigators hope to learn more about the way drugs are metabolized by pregnant women, and how those drugs are distributed in the blood and body compartments and cleared in the urine, and how maternal body weight affects the metabolism. With this information the investigators will be able to develop a treatment regimen considering factors in the body that affect magnesium levels so that the investigators can improve treatment of pregnant women. The goal of the study is to understand how different dosing of magnesium sulfate affects blood levels of the magnesium in larger women.

Magnesium sulfate is generally given to patients to protect the mother against seizures in the case of preeclampsia. Different hospitals in the United States use different doses of magnesium sulfate. Participants will receive one of two accepted doses of magnesium sulfate for preeclampsia. The dose is usually 4g - 6g at the start, with another dose of 2-3 g every hour until 24 hours after delivery. Participants will be assigned to either a dose of 4 g at the start, followed by 1g every hour; or a dose of 6 g at the start, followed by 2g every hour until treatment for preeclampsia is complete. Participants will receive magnesium sulfate in the course of their normal clinical care whether or not they participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are ages 18-45
* 32-42 weeks' pregnant
* Prescribed magnesium sulfate for preeclampsia
* BMI ≥35 kg/m2

Exclusion Criteria:

* Pregnant women < 32 weeks' pregnant
* Women who are on dialysis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Brookfield, M.D., PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science Univerity, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037
- [Derived] Brookfield KF, Tuel K, Rincon M, Vinson A, Caughey AB, Carvalho B. Alternate Dosing Protocol for Magnesium Sulfate in Obese Women With Preeclampsia: A Randomized Controlled Trial. Obstet Gynecol. 2020 Dec;136(6):1190-1194. doi: 10.1097/AOG.0000000000004137. PMID 33156201

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 66 Women were consented, enrolled and assigned a study arm for this study. However, this was prior to clinical need for intervention, therefore several women who were enrolled in the study did not show clinical need for intervention.
Groups:
- MgSO4 4g Load, 1g/hr Infusion: Once their obstetrician prescribes magnesium sulfate, participant will be assigned by 50/50 chance to one of two treatment regimens. Participant will be assigned to either a dose of 4 g at the start, followed by 1g every hour; or a dose of 6 g at the start, followed by 2g every hour until treatment for preeclampsia is complete.
  Magnesium sulfate 4g loading dose, 1g/hr infusion
- MgSO4 6g Load, 2g/hr Infusion: Once their obstetrician prescribes magnesium sulfate, participant will be assigned by 50/50 chance to one of two treatment regimens. Participant will be assigned to either a dose of 4 g at the start, followed by 1g every hour; or a dose of 6 g at the start, followed by 2g every hour until treatment for preeclampsia is complete.
  Magnesium sulfate 6g loading dose, 2g/hr infusion
Period: Overall Study
Arm/Group | MgSO4 4g Load, 1g/hr Infusion | MgSO4 6g Load, 2g/hr Infusion
Started | 31 | 35
Completed | 18 | 19
Not Completed | 13 | 16
Not completed — Did not receive allocated intervention | 13 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MgSO4 4g Load, 1g/hr Infusion | MgSO4 6g Load, 2g/hr Infusion | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.9 (6.6) | 31.6 (7.1) | 31.3 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 15 | 15 | 30
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37
BMI [Median (Inter-Quartile Range); unit: Kg/m^2] | 41 [37 to 46] | 42 [37 to 45] | 41 [37 to 46]
Multiparity [Count of Participants; unit: Participants] | 11 | 11 | 22
Baseline Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 0.6 [0.56 to 0.65] | 0.67 [0.54 to 0.73] | 0.6 [0.54 to 0.7]
Time to delivery [Median (Inter-Quartile Range); unit: Hours] | 14.7 [10.3 to 27.2] | 22.0 [13.1 to 39.0] | 19.3 [10.8 to 24.2]

OUTCOME MEASURES:

1. Primary Outcome: Maternal Serum Magnesium Level at 4 Hours After Administration
Description: magnesium level in mg/dL
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MgSO4 4g Load, 1g/hr Infusion | MgSO4 6g Load, 2g/hr Infusion
Number analyzed (Participants) | 18 | 19
mg/dL | 3.53 (.3) | 4.41 (.5)

2. Secondary Outcome: Maternal Serum Magnesium Level at Time of Delivery
Description: magnesium level in mg/dL
Time Frame: Within 20 minutes of delivery
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MgSO4 4g Load, 1g/hr Infusion | MgSO4 6g Load, 2g/hr Infusion
Number analyzed (Participants) | 18 | 19
mg/dL | 3.73 (0.7) | 5.44 (1.0)

3. Secondary Outcome: Maternal Side Effects
Description: Presence or absence of the following: flushing, lethargy, palpitations, pain at IV site, respiratory depression
Time Frame: 4 hours
Measure: Number; unit: percentage of participants
Arm/Group | MgSO4 4g Load, 1g/hr Infusion | MgSO4 6g Load, 2g/hr Infusion
Number analyzed (Participants) | 18 | 19
percentage of participants
  Nausea | 5.5 | 10.5
  Flushing | 0 | 5.2
  Lethargy | 0 | 0
  Palpitations | 0 | 0
  Pain at IV site | 0 | 0
  Respiratory depression | 0 | 0

ADVERSE EVENTS:
Time Frame: 19 months
Arm/Group | MgSO4 4g Load, 1g/hr Infusion | MgSO4 6g Load, 2g/hr Infusion
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT02835339/Prot_SAP_000.pdf